CLINICAL TRIAL: NCT05580822
Title: Additive Effects of Intra-arterial Tenecteplase for Successful Thrombectomy Due to Acute Basilar Artery Occlusion (ARTERIAL TNK BAO)：a Prospective, Randomized, Open-label, Blinded Endpoint, Multicenter, Phase 2 Study
Brief Title: Additive Effects of Intra-arterial Tenecteplase for Successful Thrombectomy Due to Acute Basilar Artery Occlusion
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Hospital of China Medical University (Other)
Responsible Party: Principal Investigator, Chuansheng Zhao, Professor, First Hospital of China Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ARTERIAL-TNK-BAO-202201
Record Dates: First submitted 2022-10-12; First posted 2022-10-14 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Basilar Artery Occlusion; Thrombectomy; Tenecteplase
MeSH Terms: interventions — Tenecteplase; Injections; Sodium Chloride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- intra-arterial TNK infusion (0.4mg/min) via support/access catheter, over 15 minutes (Experimental)
  Interventions: Drug: Tenecteplase for Injection
- intra-arterial TNK infusion (0.25mg/min) via support/access catheter, over 15 minutes (Experimental)
  Interventions: Drug: Tenecteplase for Injection
- intra-arterial placebo infusion via support/access catheter, over 15 minutes (Placebo Comparator)
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Tenecteplase for Injection — intra-arterial TNK infusing after successful thrombectomy for patient with acute basilar artery occlusion via support/access catheter
  Arms: intra-arterial TNK infusion (0.25mg/min) via support/access catheter, over 15 minutes; intra-arterial TNK infusion (0.4mg/min) via support/access catheter, over 15 minutes
Drug: Saline — intra-arterial saline infusing after successful thrombectomy for patient with acute basilar artery occlusion via support/access catheter
  Arms: intra-arterial placebo infusion via support/access catheter, over 15 minutes

SUMMARY:
Recent studies revealed the safety and effectiveness of EVT in patients with acute occlusion at basilar artery, showing that up to 46% of patients receiving EVT had favorable functional outcome at 3 months (ATTENTION and BAOCHE trials, ESOC). Although the rate of successful recanalization can be as high as 90% , a large number of these patients remains to be functionally independent while recovery. In addition, a number of recent studies indicated the functional outcome of patients with successful recanalization of TICI 2b was not as good as those with TICI 3 grade. Therefore, restoring reperfusion of distal vessels and territorial microcirculation may be pivotal to further improvement of neurological outcomes for AIS patients receiving EVT. Correspondingly, a very recent Spanish multicenter randomized trial showed the effect of further functional improvement of post-EVT intra-arterial alteplase for successful mechanical thrombectomy in anterior circulation More importantly, head-to-head comparison between TNK and tPA showed the former has a significantly higher chance of reperfusion, indicating that TNK may be a potentially better candidate for post-EVT bridging.

Based on the above findings, we hypothesize in the present study that, adjunct intra-arterial tenecteplase after successful thrombectomy could enhance the functional improvement in patients with acute basilar artery occlusion.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 - 80 yro；
2. Acute symptomatic basilar artery occlusion identified by neuroimaging modalities (CTA/MRA/DSA)；
3. NIHSS ≥ 6 before thrombectomy；
4. Time from symptom onset (or last seen normal) to arterial TNK/placebo is less than 24 hours；
5. pc-ASPECTS ≥ 6 and Pons-midbrain-index ≤ 2
6. Successful recanalization（eTICI 2b-3）at the end of procedure（The maximum will be six passes or six aspirations for the patient）；Patients with an eTICI score 2b/3 on the diagnostic cerebral angiography before the onset of MT are also eligible for the study.
7. Exclusion of parenchymal hemorrhagic transformation (DynaCT/XpertCT) before intra-arterial agent administration；
8. Pre-morbid mRS ≤ 1；
9. Patient or legal proxy is able to understand and willing to provide written inform and consent.

Exclusion Criteria:

1. Patient received thrombolysis prior to EVT
2. NIHSS score on admission >25
3. Contraindication to IA TNK as per local national guidelines (except time to therapy)
4. Use of stents during the endovascular procedure requiring dual antiplatelet therapy during the first 24h
5. Female who is pregnant or lactating or has a positive pregnancy test at time of admission
6. Current participation in another investigation drug or device treatment study (except observational study)
7. Known hereditary or acquired hemorrhagic diathesis, coagulation factor deficiency
8. Known coagulopathy, INR >1.7 or use of novel anticoagulants < 48h from symptom onset
9. Platelets <100,000
10. Renal Failure as defined by a serum creatinine >3.0 mg/dl (or 265.2 μmol/l) or glomerular Filtration Rate [GFR] <30.
11. Subject who requires hemodialysis or peritoneal dialysis, or who have a contraindication to an angiogram for whatever reason
12. Any hemorrhage on CT/MRI
13. Clinical presentation suggests a subarachnoid hemorrhage, even if initial CT or MRI scan is normal
14. Suspicion of aortic dissection
15. Subject currently uses or has a recent history of illicit drug(s) or abuses alcohol
16. History of life threatening allergy (more than rash) to TNK or contrast medium
17. SBP >185 mmHg or DBP >110 mmHg refractory to treatment
18. Serious, advanced, terminal illness with anticipated life expectancy <6 months
19. Pre-existing neurological or psychiatric disease that would confound evaluation
20. Presumed vasculitis or septic embolization
21. Unlikely to be available for 90-day follow-up (e.g. no fixed home address, visitor from overseas)
22. Other conditions at investigators' discretion which are not appropriate for participation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
mRS 0-3 | 90 days
  The proportion of patients with a modified Rankin Scale 0 to 3 at 90 days
symptomatic ICH | 24 hours
  The proportion of symptomatic ICH within 24 hours after allocated intervention

SECONDARY OUTCOMES:
mRS 0-1 | 90 days
  The proportion of patients with a mRS 0 to 1 at 90 days
mRS 0-2 | 90 days
  The proportion of patients with a mRS 0 to 2 at 90 days
mRS shift | 90 days
  The proportion of patients with a mRS shift at 90 days
early neurological improvement | 48 hours
  The proportion of patients with early neurological improvement (NIHSS reduction > 4) at 48 hours
PH1 and PH2 sICH | 24 hours
  The proportion of subtypes (PH1 and PH2) of sICH within 24 hours after allocated intervention
mortality | 90 days
  The proportion of mortality at 90 days